CLINICAL TRIAL: NCT00143819
Title: Double-Blind, Bilateral, Vehicle-Controlled, Randomized Trial of Neuroskin Forte to Relieve Symptoms of Dry Skin
Brief Title: Neuroskin Forte for Dry Skin Relief in Eczema and Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: AVVAA World Healthcare Products, Inc. (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5494
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis; Eczema
Keywords: psoriasis; dry skin; eczema; atopic dermatitis
MeSH Terms: conditions — Psoriasis; Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): bilateral comparison
  Interventions: Drug: Neuroskin Forte
- 2 (Placebo Comparator): bilateral comparison
  Interventions: Drug: Placebo Application

INTERVENTIONS:
Drug: Neuroskin Forte — Subjects will apply study drug sprays 3 times a day (with optional 4th application) to the assigned, randomized sides of the body for 8 weeks
  Arms: 1
Drug: Placebo Application — Subjects will apply placebo sprays 3 times a day (with optional 4th application) to the assigned, randomized sides of the body for 8 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of Neuroskin Forte in relieving the symptoms of dry skin in adults with psoriasis or eczema.

DETAILED DESCRIPTION:
Subjects will apply study drug and placebo sprays 3 times a day to the assigned, randomized sides of the body. They are allowed to continue using prescription medications, but not moisturizers. Assessments will be performed every other week. Total duration of the study is 10 weeks (8 weeks of treatment and a follow-up visit 2 weeks later).

ELIGIBILITY:
Inclusion Criteria

* Must be at least 18 years of age
* Have psoriasis or eczema on both sides of the body, with a pair of roughly symmetrical bilateral "target" lesions at least 1.5 cm in diameter

Exclusion Criteria

* Inability to understand the consent form and/or comply with the requirements of this study
* Use of moisturizers/emollients within 2 days of beginning study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Magliocco, MD, Principal Investigator — Rutgers, The State University of New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 (Left Side: Active; Right Side: Placebo): bilateral comparison
  Subjects randomized to Group 1 applied Neuroskin Forte study drug sprays to the left side of the body and placebo sprays to the right side of the body, 3 times a day (with optional 4th application), for 8 weeks.
- 2 (Left Side: Placebo; Right Side: Active): bilateral comparison
  Subjects randomized to Group 2 applied placebo sprays to the left side of the body and Neuroskin Forte study drug sprays to the right side of the body, 3 times a day (with optional 4th application), for 8 weeks.
Period: Overall Study
Arm/Group | 1 (Left Side: Active; Right Side: Placebo) | 2 (Left Side: Placebo; Right Side: Active)
Started | 5 | 8
Completed | 3 | 5
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Bilateral Comparison Group 1: bilateral comparison
  Neuroskin Forte: Subjects will apply study drug sprays 3 times a day (with optional 4th application) to the assigned, randomized sides of the body for 8 weeks
- Bilateral Comparison Group 2: bilateral comparison
  Placebo Application: Subjects will apply placebo sprays 3 times a day (with optional 4th application) to the assigned, randomized sides of the body for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Bilateral Comparison Group 1 | Bilateral Comparison Group 2 | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 66 [49 to 79] | 61 [42 to 85] | 63 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Visual Analog Scale (VAS) Score for Pruritus (Itching) at 8 Weeks
Description: Subjects assessed the level of pruritus (itching) on the left and right sides of their body at each visit, ticking the values on a 100-mm scale (0 mm = no itching; 100 mm = worst possible itching) for each side. Percent change from baseline was calculated.
Time Frame: 8 weeks
Population: Thirteen (13) subjects were randomized to receive Neuroskin Forte (ie, active) spray on one side of the body and placebo spray on the other side of the body.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Neuroskin Forte Spray: bilateral comparison
  Subjects were randomized to apply Neuroskin Forte study drug spray to one side of the body 3 times a day (with optional 4th application), for 8 weeks.
- Placebo Spray: bilateral comparison
  Subjects were randomized to apply placebo spray to one side of the body, 3 times a day (with optional 4th application), for 8 weeks.
Arm/Group | Neuroskin Forte Spray | Placebo Spray
Number analyzed (Participants) | 13 | 13
percent change | -52.2 (34.6) | -36.2 (28.5)

2. Secondary Outcome: Number of Participants With a Psoriasis ½-Body Physician Global Assessment (PGA) Improvement of at Least 2 Levels
Description: For subjects with psoriasis, a global assessment (scale of 0-5: 0 = clear except for residual discoloration; 1 = minimal; 2 = mild; 3 = moderate; 4 = marked; 5 = severe) was performed and a score recorded for each side of the subject's body, at each visit.
Time Frame: 8 weeks
Population: The eight (8) subjects in the study who had psoriasis were randomized to receive Neuroskin Forte (ie, active) spray on one side of the body and placebo spray on the other side of the body.
Measure: Count of Participants; unit: Participants
Groups:
- Neuroskin Forte Spray (Psoriasis Patients): bilateral comparison
  Subjects were randomized to apply Neuroskin Forte study drug spray to one side of the body 3 times a day (with optional 4th application), for 8 weeks.
- Placebo Spray (Psoriasis Patients): bilateral comparison
  Subjects were randomized to apply placebo spray to one side of the body 3 times a day (with optional 4th application), for 8 weeks.
Arm/Group | Neuroskin Forte Spray (Psoriasis Patients) | Placebo Spray (Psoriasis Patients)
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With an Eczema ½-Body Investigator Global Assessment (IGA) Improvement of at Least 2 Levels
Description: For subjects with eczema, a global assessment (scale of 0-5: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe; 5 = very severe) was performed and a score recorded for each side of the subject's body, at each visit.
Time Frame: 8 weeks
Population: The five (5) subjects in the study who had eczema were randomized to receive Neuroskin Forte (ie, active) spray on one side of the body and placebo spray on the other side of the body.
Measure: Count of Participants; unit: Participants
Groups:
- Neuroskin Forte Spray (Eczema Patients): bilateral comparison
  Subjects were randomized to apply Neuroskin Forte study drug spray to one side of the body 3 times a day (with optional 4th application), for 8 weeks.
- Placebo Spray (Eczema Patients): bilateral comparison
  Subjects were randomized to apply placebo spray to one side of the body, 3 times a day (with optional 4th application), for 8 weeks.
Arm/Group | Neuroskin Forte Spray (Eczema Patients) | Placebo Spray (Eczema Patients)
Number analyzed (Participants) | 5 | 5
Participants | 1 | 0

4. Secondary Outcome: Change in Target Lesion Scoring
Description: The subjects' target lesions (ie, a pair of roughly symmetrical bilateral lesions) on each side of the body were scored by the investigator at each visit. Percent change from baseline was calculated.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo Spray: bilateral comparison
  Subjects were randomized to apply placebo spray to one side of the body 3 times a day (with optional 4th application), for 8 weeks.
Arm/Group | Neuroskin Forte Spray | Placebo Spray
Number analyzed (Participants) | 13 | 13
percent change | -20.7 (27.5) | -14.7 (11.7)

5. Secondary Outcome: Photography of Target Lesions
Description: Number of participants with photographs taken
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroskin Forte Spray | Placebo Spray
Number analyzed (Participants) | 13 | 13
Participants | 13 | 13

ADVERSE EVENTS:
Groups:
- Bilateral Comparison: Neuroskin Forte Spray vs Placebo Spray: bilateral comparison
  Subjects were randomized to apply Neuroskin Forte study drug spray to one side of the body and placebo spray to the other side of the body, 3 times a day (with optional 4th application), for 8 weeks.
Arm/Group | Bilateral Comparison: Neuroskin Forte Spray vs Placebo Spray
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral Comparison: Neuroskin Forte Spray vs Placebo Spray (N=13)
skin infection (Infections and infestations) | 1 (1)
increased itching (Skin and subcutaneous tissue disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
increased severity of eczema (Skin and subcutaneous tissue disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No